CLINICAL TRIAL: NCT06131021
Title: Shaping the Indications for Periodontal Adjunctive Antibiotics in Dental Practice: A PBRN Clinical Trial
Brief Title: Shaping the Indications for Periodontal Adjunctive Antibiotics in Dental Practice
Acronym: PAAS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH); National Dental PBRN (Unknown)
Responsible Party: Principal Investigator, Georgios A. Kotsakis, DDS, MS, Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro2023001347; 4UH3DE031129-02 (NIH)
Record Dates: First submitted 2023-10-31; First posted 2023-11-14 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Periodontitis; Periodontal Diseases; Periodontal Pocket
Keywords: Antibiotics; Amoxicillin; Metronidazole
MeSH Terms: conditions — Periodontitis; Periodontal Diseases; Periodontal Pocket | interventions — Amoxicillin; Metronidazole

STUDY DESIGN:
Intervention Model Description: The sample size will be a target of approximately 150 patient participants enrolled from up to 34 National Dental PBRN practices. All patient participants are indicated to receive SRP and have been diagnosed with periodontitis stages II-III, grades A-C. A double-blinded patient participant-randomized design is used to assign patient participants to SRP plus AMXM versus SRP plus placebo prior to treatment.
Who Masked: Participant, Care Provider
Masking Description: PBRN practitioner- and patient participant-level masking. Statistician assessor will also remain blinded; a separate biostatistician will remain unblinded in order to implement randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test Arm (Experimental): Patient participants in this arm will receive a combination of Amoxicillin 500mg & Metronidazole 500mg orally (AMXM) as adjuncts along with their scheduled non-surgical periodontal treatment as the study intervention. A loading dose of 1g of Amoxicillin and 1g of Metronidazole will be given 30-60 minutes prior to periodontal treatment. After the loading dose, each patient participant will be instructed to take Amoxicillin 500mg & Metronidazole 500mg every 8 hours for 10 days.
  Interventions: Drug: Amoxicillin; Drug: Metronidazole
- Control Arm (Placebo Comparator): Patient participants in this arm will receive a placebo capsules identical to the study drug capsules along with their scheduled non-surgical periodontal treatment as the placebo comparator in an identical frequency and duration fashion as the active drug group.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Amoxicillin — Amoxicillin belongs to the penicillin category, and it is a commonly prescribed broad-spectrum antibiotic as a periodontal treatment adjunct.
  Arms: Test Arm
Drug: Metronidazole — Metronidazole is effective against anaerobic bacteria, and it is often combined with Amoxicillin for an enhanced antimicrobial effect as a periodontal treatment adjunct.
  Arms: Test Arm
Other: Placebo — Placebo in identical drug-safe vials with capsules identical in appearance to the active drugs
  Arms: Control Arm

SUMMARY:
Periodontitis is a bacterial inflammatory disease and antibiotic use is being empirically used as part of its treatment. However, a clinical practice guideline on periodontal treatment adjuncts published in 2015 identified weak evidence on the use of systemic antibiotics and large heterogeneity across small scale studies, suggesting that larger pragmatic clinical trials would benefit clinical decision making. This will be a prospective, randomized, placebo-controlled trial, stratified by practice and practitioner. The study will investigate the effectiveness of adjunctive antibiotics as adjunct to scaling and root planing (SRP) compared to SRP with placebo for the treatment of generalized stage II-III, grades A-C periodontitis in patient participants from National Dental PBRN practices. Periodontal data will be collected at baseline, re-evaluation (6 weeks), and final (4-12 months) study visits. Changes in periodontal clinical and patient-reported outcomes will be assessed to determine the effectiveness of SRP plus adjunctive systemic Amoxicillin / Metronidazole antibiotics (AMXM) versus SRP with Placebo.

DETAILED DESCRIPTION:
Précis: Periodontitis is a bacterial inflammatory disease and antibiotic use is being empirically used as part of its treatment. However, a clinical practice guideline on periodontal treatment adjuncts published in 2015 identified weak evidence on the use of systemic antibiotics and large heterogeneity across small scale studies, suggesting that larger pragmatic clinical trials would benefit clinical decision making. This will be a prospective, randomized, placebo-controlled trial, stratified by practice and practitioner. The study will investigate the effectiveness of adjunctive antibiotics as adjunct to scaling and root planing (SRP) compared to SRP with placebo for the treatment of generalized stage II-III, grades A-C periodontitis in patient participants from National Dental PBRN practices. Periodontal data will be collected at baseline, re-evaluation (6 weeks), and final (4-12 months) study visits. Changes in periodontal clinical and patient-reported outcomes will be assessed to determine the effectiveness of SRP plus adjunctive systemic Amoxicillin / Metronidazole antibiotics (AMXM) versus SRP with Placebo.

Objectives and Outcomes: Primary: The primary objective will assess the effectiveness of SRP plus adjunctive antibiotics compared to SRP with placebo in periodontitis individuals from baseline to 6 weeks following non-surgical periodontal therapy (NSPT) as determined by changes in site-level periodontal probing depth (PD).

Secondary: To assess changes in: i) gingival inflammation (measured by bleeding on probing (BoP)), ii) periodontal tissue attachment (measured by clinical attachment level (CAL)), iii) reduction in diseased sites (measured by remaining sites with maximum probing depth ≥5 mm), and iv) disease remission (measured by number of participants with ≤4 sites with PD≥ 5mm); comparing SRP plus AMXM to SRP with a placebo adjunctive in periodontitis individuals from baseline to re-evaluation (6 weeks) to final (12 month) study visit following intervention. Also, assess changes in periodontal probing depth from baseline measurements to final visit (4-12 months) following intervention. The patient-reported impact of periodontal treatment (measured by the Oral Health Impact Profile-5 (OHIP-5)) and treatment-related adverse events between groups will also be assessed.

Population: A sample size of 150 patient participants enrolled from up to 34 National Dental PBRN practices will be enrolled for adequate power. All patient participants are indicated to receive SRP and have been diagnosed with periodontitis stages II-III, grades A-C.

Description of Intervention: The intervention will involve either SRP, which is considered the standard of care treatment for debriding root surfaces, in conjunction with 500 mg Amoxicillin and 500mg Metronidazole orally every 8 hours (q8h) for ten days following SRP or SRP with placebo.

ELIGIBILITY:
Inclusion Criteria:

* The study will recruit patient participants presenting for periodontal treatment within the National Dental PBRN practices participating in this study.

To be eligible to participate in this study, a potential patient participant must meet all the following criteria:

* Adult who is at least 35 years old.
* Presence of ≥ 15 permanent teeth excluding 3rd molars.
* In good general health as evidenced by medical history (ASA Class I or II) per the practitioner.
* Planned to receive periodontal care for Generalized Periodontitis and a minimum of two quadrants of SRP (CDT code 4341) in practices participating in the National Dental PBRN.
* Willing to comply with all study visits and be available for the duration of the study (12-15 months)
* Willing to provide contact information for self, including a cellular phone number for study text, and one to two emergency contacts to be reached for the follow-up visits and any other study-related matters for the duration of the study.

Exclusion Criteria:

* Known drug allergy to any antibiotics or anesthetics.
* Use of systemic antibiotics taken within the previous 3 months prior to enrollment.
* Medical condition which requires antibiotic prophylaxis prior to dental treatments/visits.
* Current use of medications that, in the opinion of the practitioner, may cause adverse effects with AMXM (such as disulfiram, warfarin, and oral contraceptives).
* History of any periodontal therapy (including SRP D4341, D4342) within the last 6 months prior to enrollment.
* Is currently pregnant or lactating per patient participant self-report.
* Is considered immunocompromised, in the opinion of the practitioner (including diseases and conditions such as HIV/AIDS, immunosuppressive drug therapy and/or radiation), or has chronic mucosal lesions (e.g. pemphigus vulgaris) affecting the gingiva.
* Has Diabetes mellitus with an HbA1c score of >/= 10% within the past 3 months as per patient participant self-report.

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-04-25 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-05-26 (Estimated)

PRIMARY OUTCOMES:
Probing Depth (PD) in millimeters | Baseline to Re-evaluation (6 weeks)
  The primary outcome of treatment effectiveness will be assessed by full-mouth probing depth (PD) from baseline to 6 weeks following intervention. Full-mouth PD measurements (excluding 3rd molars) will be obtained utilizing a UNC 15mm periodontal probe.

SECONDARY OUTCOMES:
Clinical attachment level (CAL) in millimeters | Baseline, Re-evaluation (6 weeks), and Final study visit (12 months) after intervention.
  This secondary objective will be assessed by clinical attachment level (CAL) changes from baseline to 6 weeks to 12 months post-intervention, adjusting for baseline CAL. CAL is a disease-related characteristic. Half-mouth CAL in millimeters (excluding 3rd molars) will be obtained utilizing a UNC 15mm periodontal probe to measure base of pocket to cementoenamel junction (CEJ).
Changes in the probability of bleeding on probing (BoP) | Baseline, Re-evaluation (6 weeks), and Final study visit (12 months) after intervention.
  This secondary objective will assess changes in the probability of observing BoP, a common surrogate for gingival inflammation, at 6 weeks to 12 months post intervention, adjusting for baseline BoP. BoP is assessed in conjunction with probing depths using a UNC 15mm periodontal probe and is recorded as a binary outcome per site, i.e., is the site bleeding? Yes/No.
Reduction in diseased sites | Baseline, Re-evaluation (6 weeks), and Final study visit (12 months) after intervention.
  Reduction in diseased sites is a calculated variable from PD. We will assess the probability a site is observed with residual PD≥ 5 mm at 6 weeks to 12 months post-intervention, adjusting for its baseline PD. PD≥ 5mm; The maximum probing depth per tooth will be recorded as ≥5 mm (yes/no).
Disease remission | Baseline, Re-evaluation (6 weeks), and Final study visit (12 months) after intervention.
  Disease remission is defined as the number of study patient participants who have ≤4 sites with PD≥5mm. Patient participants will be considered 'in remission' if they display ≤4 sites with PD≥ 5mm; This is a dichotomization from the summation of PD≥ 5mm within person.
Changes in oral health-related quality of life | Baseline, Re-evaluation (6 weeks), and Final study visit (12 months) after intervention.
  To evaluate oral health-related quality of life, the Oral Health Impact Profile (OHIP-5) will be utilized. OHIP-5 sum score based upon self-reported responses will be assessed. The OHIP-5 has 5 questions ranging from 0 = never to 4 = very often with higher scores translating to a worse outcome.
Probing Depth (PD) in millimeters at final visit | Baseline, Final study visit (4-12 months) after intervention.
  This secondary outcome of treatment effectiveness will be assessed by the change in full-mouth probing depth (PD) from baseline to 4-12 months post-intervention. Full-mouth PD measurements (excluding 3rd molars) will be obtained utilizing a UNC 15mm periodontal probe.

OTHER OUTCOMES:
Treatment-related adverse events | Through study completion, an average of 12 months
  The number and severity of adverse events related to SRP plus AMXM versus SRP plus placebo will be recorded to assess the safety of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Georgios Kotsakis, DDS, Principal Investigator — Rutgers University
Locations (1):
- University of Alabame, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.nationaldentalpbrn.org/blog/paas/